CLINICAL TRIAL: NCT07145879
Title: Differences in Soft Tissue Healing and Vascularization Between Articaine and Lidocaine: A Randomized Clinical and Ultrasonographic Study
Brief Title: Comparison of Postoperative Effects of Articaine and Lidocaine in Mucogingival Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, AYSAN LEKTEMUR ALPAN, Head of Periodontology Department, Pamukkale University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Diagnostic
Other Study IDs: 07.01.2025/01
Record Dates: First submitted 2025-08-14; First posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Local Analgesia Via Infiltration; Wound Heal; Pain, Postoperative; Hemorrhage
Keywords: wound healing; free gingival graft; pain; dental anxiety; local anaesthesia
MeSH Terms: conditions — Pain, Postoperative; Hemorrhage; Pain | interventions — Lidocaine; Epinephrine; Carticaine

STUDY DESIGN:
Intervention Model Description: prospective cross sectional study
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- lidocaine HCL (Other): Participants will receive lidocaine HCL 2% with adrenaline for local anesthesia before free gingival surgery once only
  Interventions: Drug: Lidocaine hydrochloride 2% with epinephrine 1:100 000; Procedure: Free gingival graft (FGG)
- articaine HCL (Other): Participants will receive articaine HCL 4% with adrenaline for local anestesia before free gingival surgery once only
  Interventions: Drug: Articaine 4% with epinephrine 1:100,000; Procedure: Free gingival graft (FGG)

INTERVENTIONS:
Drug: Lidocaine hydrochloride 2% with epinephrine 1:100 000 — Patient were received infiltrative anesthesia with Lidocaine (Jetokain, Adeka Ilaç, Samsun, Türkiye): Active ingredient: Each 1 ml contains 20 mg lidocaine hydrochloride (HCL) and 0.012 mg epinephrine base. Excipients: Sodium metabisulfite, sodium chloride, water for injection.
  Other Names: free gingival graft
  Arms: lidocaine HCL
Drug: Articaine 4% with epinephrine 1:100,000 — Patients were received Infiltrative anesthesia with Articaine (Ultracain DS Forte, Sanofi Aventis İlaçları, Istanbul, Türkiye): Active ingredient: 40 mg articaine HCL and 0.012 mg epinephrine per 1 ml. Excipients: Sodium chloride, sodium metabisulfite, hydrochloric acid, water for injection
  Other Names: free gingival graft
  Arms: articaine HCL
Procedure: Free gingival graft (FGG) — FGG surgery was performed around natural teeth and implants where keratinized gingival tissue was inadequate.

SUMMARY:
The aim of this study is to compare and evaluate the effects of using lidocaine 2% (with adrenaline) and articaine 4% (with adrenaline) in free gingival graft (FGG) surgery on postoperative wound healing, changes in blood flow in the surgical area during the healing process, patients' postoperative pain levels, and anxiety levels before and after surgery.

DETAILED DESCRIPTION:
In a prospective randomised controlled trial conducted to investigate the effect of lidocaine and articaine on postoperative free gingival graft healing, wound healing was assessed using EHS, anxiety was assessed using VAS, STAI, and MDAS questionnaires, and ultrasonographic evaluations and PI measurements were used to determine whether there was a difference in wound healing between the two anaesthetics.

ELIGIBILITY:
Inclusion Criteria:

* Patients> 18 years requiring FGG surgery with ≤ 1 mm width of attached gingiva
* No systemic diseases or pregnancy.
* Smoking ≤10 cigarettes/day
* Full-mouth plaque score and full-mouth bleeding score ≤10% (four sites per tooth).
* Need for FGG due to insufficient attached gingiva
* No history of mucogingival or periodontal surgery at experimental sites

Exclusion Criteria:

* Use of oral contraceptives, psychotropic drugs, sedatives, or NSAIDs
* Allergy or hypersensitivity to local anesthetics,
* Orofacial neurological symptoms,
* Active infection in the surgical area,
* Pathological mental conditions such as dementia or psychosis, or lack of cooperation,

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
early wound healing score (EHS) | 3rd day, 7th day, 14th day
  The healing of the recipient site was evaluated using the EHS index during clinical exams on postoperative days 3, 7, and 14. The EHS index includes parameters of hemostasis (CSH), inflammation (CSI), and re-epithelialization (CSR). The total score ranges from 0 (worst healing) to 10 (best healing)

SECONDARY OUTCOMES:
Ultrasonographic Evaluations | 3rd, 7th, and 14th days
  All patients were evaluated using an ultrasonography (USG) device (MyLab™ Seven, Esaote, Genoa, Italy) in the Department of Oral and Maxillofacial Radiology. USG examinations were performed by an oral and maxillofacial radiologist with at least eight years of experience before graft harvesting and on the 3rd, 7th, and 14th days after FGG operations in both recipient and donor sites.
Modified Dental Anxiety Scale (MDAS) | baseline and 14 days after the procedure,
  The MDAS includes five scores that progressively increase from "not anxious" to "extremely anxious" for each question. Therefore, the highest score for each question is 5, and the total score for the scale ranges from 5 to 25, with 25 being the maximum
State-Trait Anxiety Inventory (STAI-S and STAI-T) | baseline and 14 days after the procedure,
  The trait anxiety section (STAI-T) helps measure how the individual has felt over the past weeks, while the state anxiety section (STAI-S) is designed to assess how the individual feels at that moment. Participants are asked to select the statement that best describes their feelings from the options provided: "definitely not," "sometimes," "often," or "almost always." Positive scores were assigned to the statements in items 3, 4, 6, 7, 9, 12, 13, 14, 17, and 18, while negative scores were assigned to the statements in items 1, 2, 5, 8, 10, 11, 15, 16, 19, and 20. A score of 80 was considered the highest, while 20 was the lowest

CONTACTS AND LOCATIONS:
Overall Officials: Aysan Lektemur Alpan, PhD DDS, Principal Investigator — Pamukkale University Faculty of Dentistry
Locations (1):
- Pamukkale University Faculty of Dentistry, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I can share it after my article is published if there is a valid reason.

REFERENCES:
- [Background] Kesici S, Kesici U, Ulusoy H, Erturkuner P, Turkmen A, Arda O. [Effects of local anesthetics on wound healing]. Braz J Anesthesiol. 2018 Jul-Aug;68(4):375-382. doi: 10.1016/j.bjan.2018.01.016. Epub 2018 Jun 6. PMID 29884529
- [Background] Al-Saffar, M.T., A.S. Mahmood, and M.S. Sulaiman, Impact of Local Anesthesia on Wound Healing. Indian Journal of Forensic Medicine & Toxicology, 2020. 14(4): p. 1869-1874.
- [Background] Giovannitti JA Jr, Rosenberg MB, Phero JC. Pharmacology of local anesthetics used in oral surgery. Oral Maxillofac Surg Clin North Am. 2013 Aug;25(3):453-65, vi. doi: 10.1016/j.coms.2013.03.003. Epub 2013 May 7. PMID 23660127
- [Background] Luo W, Zheng K, Kuang H, Li Z, Wang J, Mei J. The potential of articaine as new generation of local anesthesia in dental clinics: A review. Medicine (Baltimore). 2022 Dec 2;101(48):e32089. doi: 10.1097/MD.0000000000032089. PMID 36482533